CLINICAL TRIAL: NCT01157533
Title: Utility of Vancomycin Loading: A Pharmacokinetic Analysis in Critically Ill Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0887
Record Dates: First submitted 2010-07-05; First posted 2010-07-07 (Estimated); Results first posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-02

CONDITIONS: Infection
Keywords: Vancomycin; Pharmacokinetic testing; PK
MeSH Terms: conditions — Infections | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vancomycin Loading (Experimental): Loading dose 30 mg/kg via central or peripheral intravenous infusion. Subsequent doses of vancomycin (15 mg/kg) are considered standard of care.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Loading dose 30 mg/kg via central or peripheral intravenous infusion. Subsequent doses of vancomycin (15 mg/kg) are considered standard of care.

SUMMARY:
The goal of this clinical research study is to learn if giving a larger than normal "loading dose" of the antibiotic vancomycin before starting standard vancomycin dosing can help patients reach and maintain the needed blood-level of the antibiotic during treatment.

DETAILED DESCRIPTION:
The Study Drug:

Vancomycin is an antibiotic used to treat serious, life-threatening infections caused by bacteria. Researchers want to find the best and most effective dose and blood-level of the drug that may have the best effect against bacteria.

Study Drug Administration:

If your doctor believes you are eligible, and you agree to take part in this study, you will be given a "loading dose" of vancomycin that is about twice as large as the standard dose. The dose amounts will be based on your body weight. Doses can be given every 8-12 hours, depending on your level of kidney function.

Study Procedures:

Blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing and to check your kidney function. PK testing measures the amount of study drug in the body at different time points. PK blood samples will be drawn just after the loading dose, and then just before each standard dose of vancomycin (up to 5 samples total). When possible, the PK sample may be drawn through a central venous catheter or line you already have placed, to avoid extra "needle sticks."

The study staff will collect information about your health and any side effects you may be having for 7 days.

Length of Study:

Treatment with vancomycin may be stopped early if you experience intolerable side effects or the doctor thinks you can stop taking the drug early.

This is an investigational study. Vancomycin is FDA approved and commercially available for use in treating bacterial infection. The use of a loading dose for vancomycin is investigational.

Up to 10 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to MD Anderson Cancer Center Surgical Intensive Care Unit (SICU) under the Thoracic Surgery physician group
2. Intravenous vancomycin therapy deemed necessary

Exclusion Criteria:

1. Age less than 18 years
2. History of hypersensitivity to vancomycin
3. Patient weight greater than 150 kg
4. Receival of 1 or more doses of the following agents within 72 hours prior to screening: amphotericin B (lipid, liposomal, or conventional formulation), aminoglycosides, foscarnet and/or intravenous contrast dye.
5. Prior exposure (within 7 days) to intravenous vancomycin
6. Current renal insufficiency defined as baseline Scr >/= 1.5 mg/dL, or increase in baseline serum creatinine (SCr) by >/= 0.5 mg/dL within the last 2 days, or estimated creatinine clearance (CrCl) </= 30 mL/min by Cockcroft-Gault equation.
7. Current need for hemodialysis or continuous renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ara Vaporciyan, MD, BS, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas (UT) MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 21, 2010 to January 4, 2012. All recruitment done at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Vancomycin Loading
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vancomycin Loading
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Attaining Target Trough of 15-20 mg/L Following 30 mg/kg Loading Dose
Description: Peak level (PK blood samples) drawn 4 hours after the completion of loading dose. Sequential trough levels drawn 30 minutes before each standard vancomycin dose for the next 4 doses. PK testing measures the amount of study drug in the body at different time points, with trough testing following 5 doses (1 dose every 8 to 12 hours).
Time Frame: Up to 5 days
Population: Unable to complete analysis planned due to low enrollment.
Arm/Group | Vancomycin Loading
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Vancomycin Loading
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No